CLINICAL TRIAL: NCT06566391
Title: Primary Ipilimumab and Nivolumab Combo-immunotherapy Followed by Adjuvant Nivolumab in Locally Advanced or Limited Metastatic Melanoma
Brief Title: Ipilimumab and Nivolumab Followed by Adjuvant Nivolumab in Locally Advanced or Limited Metastatic Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO 838
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-02

CONDITIONS: Melanoma
Keywords: Locally advanced melanoma; Metastatic melanoma; Immunotherapy
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ipilimumab + Nivolumab followed by Nivolumab (Experimental): Neoadjuvant therapy: Ipilimumab 1 mg/kg + Nivolumab 3mg/kg every 3 weeks for 4 cycles; Adjuvant therapy: Nivolumab 480 mg every 4 weeks for 6 cycles
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Nivolumab and Ipilimumab (sequential) for a total of four doses followed by Nivolumab
  Other Names: Nivolumab

SUMMARY:
This is open label, single arm study for pts with stage IIIB-IV melanoma, accordingly with AJCC staging criteria (8th ed.), with potentially resectable disease. Patients will receive every three weeks, four cycles of Nivolumab 3 mg/kg (over one 30 minutes infusion) and Ipilimumab 1 mg/kg (over 30 minutes infusion) with a 30 minute break between each infusion. Surgery will be performed after 4-6 weeks from the last dose. After 4-6 weeks from surgery, patients will receive Nivolumab 480 mg (over one 60 minutes infusion), every four weeks for six cycles.

The duration of the trial is expected to be 12 months of accrual and approximately 24 months of follow-up after the end of adjuvant therapy.

DETAILED DESCRIPTION:
The study begins by establishing the patient's initial eligibility and signing of the ICF. Blood samples and tumor tissue obtained from core biopsy must be provided for biomarker analyses.

All patients will receive every three weeks cycles of combined Nivolumab 3 mg/kg and Ipilimumab 1 mg/kg (sequential) for a total of four doses. Nivolumab and Ipilimumab will be administered sequentially, as two separate infusions, one 30 minute Nivolumab infusion and one 30 minute Ipilimumab infusion with a 30 minute break between each infusion.

Surgery will be performed on Week 12-16 on known disease sites and in absence of G2-3-4 AE.

The Adjuvant treatment will be performed on Week 16-22 from surgery; it will consist in Nivolumab 480 mg (over one 60 minutes infusion), every four weeks for six cycles.

The Follow-up period will start 4 weeks after the end of adjuvant therapy. Patients will be followed for 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed 8th ed. AJCC Stage IIIB/C/D or Stage IV oligometastatic resectable melanoma. Patients with cutaneous, mucosal, acral, ocular or unknown primary melanomas are eligible for enrollment. Oligometastatic melanoma is defined as three or fewer areas of resectable disease excluding central nervous system and bone involvement. In case of involvement of three areas, one must be superficial (cutaneous-subcutaneous). Resectable tumors are defined as having no significant vascular, neural or bony involvement. A multidisciplinary discussion within surgical oncologists, medical oncologists, and radiologist will assess if disease is resectable.
2. Signed Written Informed Consent.
3. Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and all protocol procedures.
4. Males and Females, ages ≥18 years of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
6. Have measurable disease based on RECIST 1.1.
7. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion at baseline and at the time points specified in the Study Procedure Tables.
8. Known BRAF V600 mutation status as determined by local institutional standard. All BRAF statuses (BRAF wild type or BRAF 600 mutation positive) are eligible.
9. Patients who have been previously treated in the adjuvant setting for melanoma will be eligible for treatment after a 28 day washout period.
10. Patients must be medically fit enough to undergo surgery as determined by the treating medical and surgical oncology team.
11. Demonstrate adequate organ function as defined below: Hematologic Absolute neutrophil count (ANC) >/= 1.5 X 10^9/L; Hemoglobin >/= 9.5 g/dL Platelets >/= 100 X 10^9/L PT/INR and PTT </= 1.5 X ULN. Hepatic Total bilirubin </= 1.5 X ULN (isolated bilirubin >1.5 X ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) AST and ALT Albumin </= 2.5 X ULN 1 >/=2.5 g/dL Renal Creatinine OR Calculated creatinine clearance OR 24-hour urine creatinine clearance </=1.5 X ULN 2 >/= 50 mL/min >/= 50 mL/min.
12. Women are eligible to participate if: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/mL and estradiol < 40 pg/mL (<140 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT.
13. The individual methods of contraception and duration should be determined in consultation with the investigator. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product.
14. Women must not be breastfeeding.
15. Men who are sexually active must use any contraceptive method with a failure rate of less than 1% per year. The investigator shall review contraception methods and the time period that contraception must be followed.
16. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) and azoospermic men do not require contraception

Exclusion Criteria:

1. Currently receiving cancer therapy (chemotherapy, radiation therapy, immunotherapy, or biologic therapy) or investigational anti-cancer drug.
2. Any major surgery within the last 3 weeks.
3. Brain metastases, leptomeningeal disease or bone metastases.
4. Pregnant or lactating female.
5. Unwillingness or inability to follow the procedures required in the protocol.
6. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
7. Prior malignancy active within the previous 2 years except for patient's prior diagnosis of melanoma and locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast with local control measures (surgery, radiation).
8. Patients with active, known or suspected autoimmune disease. Patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
9. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
10. Prior treatment with an anti-PD-1, anti-PD-L1 or anti-CTLA-4 antibody.
11. Any positive test result for hepatitis B or C virus indicating acute or chronic infection.
12. Known history of testing positive for human immunodeficiency virus or known acquired immunodeficiency syndrome.
13. History of severe hypersensitivity reaction to any monoclonal antibody.
14. Prisoners or patients who are involuntarily incarcerated.
15. Patients who are compulsorily detained for treatment of either a psychiatric or physical (infection disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of pathological complete response (Efficacy) | 12-16 weeks after Neoadjuvant therapy
  Efficacy assessment is pathological complete remission rate, documented after neoadjuvant therapy.

SECONDARY OUTCOMES:
Rates of 3-4 AEs | 24 months
  Rates of grade 3-4 AE rates (immune related or not) of neoadjuvant and adjuvant regimen
Overall AE rates | up to 24 months after the end of adjuvant therapy
  Overall AE rates (immune related or not)
Patients completing treatment schedule. | up to 24 months after the end of adjuvant therapy
  Rates of pts completing treatment schedule.
Overall Response Rate (ORR) | 12-14 weeks
  Overall Response Rate (ORR), according to RECIST 1.1 criteria.
Overall Survival (OS) | 12-14 weeks
  Overall Survival (OS), according to RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Nezi, PhD, Principal Investigator — Istituto Europeo di Oncologia
Locations (1):
- Istituto Europeo di Oncologia, Milan, Italy

REFERENCES:
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Robert C, Long GV, Brady B, Dutriaux C, Maio M, Mortier L, Hassel JC, Rutkowski P, McNeil C, Kalinka-Warzocha E, Savage KJ, Hernberg MM, Lebbe C, Charles J, Mihalcioiu C, Chiarion-Sileni V, Mauch C, Cognetti F, Arance A, Schmidt H, Schadendorf D, Gogas H, Lundgren-Eriksson L, Horak C, Sharkey B, Waxman IM, Atkinson V, Ascierto PA. Nivolumab in previously untreated melanoma without BRAF mutation. N Engl J Med. 2015 Jan 22;372(4):320-30. doi: 10.1056/NEJMoa1412082. Epub 2014 Nov 16. PMID 25399552
- [Background] Robert C, Schachter J, Long GV, Arance A, Grob JJ, Mortier L, Daud A, Carlino MS, McNeil C, Lotem M, Larkin J, Lorigan P, Neyns B, Blank CU, Hamid O, Mateus C, Shapira-Frommer R, Kosh M, Zhou H, Ibrahim N, Ebbinghaus S, Ribas A; KEYNOTE-006 investigators. Pembrolizumab versus Ipilimumab in Advanced Melanoma. N Engl J Med. 2015 Jun 25;372(26):2521-32. doi: 10.1056/NEJMoa1503093. Epub 2015 Apr 19. PMID 25891173
- [Background] Hodi FS, Chesney J, Pavlick AC, Robert C, Grossmann KF, McDermott DF, Linette GP, Meyer N, Giguere JK, Agarwala SS, Shaheen M, Ernstoff MS, Minor DR, Salama AK, Taylor MH, Ott PA, Horak C, Gagnier P, Jiang J, Wolchok JD, Postow MA. Combined nivolumab and ipilimumab versus ipilimumab alone in patients with advanced melanoma: 2-year overall survival outcomes in a multicentre, randomised, controlled, phase 2 trial. Lancet Oncol. 2016 Nov;17(11):1558-1568. doi: 10.1016/S1470-2045(16)30366-7. Epub 2016 Sep 9. PMID 27622997
- [Background] Wolchok JD, Chiarion-Sileni V, Gonzalez R, Rutkowski P, Grob JJ, Cowey CL, Lao CD, Wagstaff J, Schadendorf D, Ferrucci PF, Smylie M, Dummer R, Hill A, Hogg D, Haanen J, Carlino MS, Bechter O, Maio M, Marquez-Rodas I, Guidoboni M, McArthur G, Lebbe C, Ascierto PA, Long GV, Cebon J, Sosman J, Postow MA, Callahan MK, Walker D, Rollin L, Bhore R, Hodi FS, Larkin J. Overall Survival with Combined Nivolumab and Ipilimumab in Advanced Melanoma. N Engl J Med. 2017 Oct 5;377(14):1345-1356. doi: 10.1056/NEJMoa1709684. Epub 2017 Sep 11. PMID 28889792
- [Background] Long GV, Atkinson V, Cebon JS, Jameson MB, Fitzharris BM, McNeil CM, Hill AG, Ribas A, Atkins MB, Thompson JA, Hwu WJ, Hodi FS, Menzies AM, Guminski AD, Kefford R, Kong BY, Tamjid B, Srivastava A, Lomax AJ, Islam M, Shu X, Ebbinghaus S, Ibrahim N, Carlino MS. Standard-dose pembrolizumab in combination with reduced-dose ipilimumab for patients with advanced melanoma (KEYNOTE-029): an open-label, phase 1b trial. Lancet Oncol. 2017 Sep;18(9):1202-1210. doi: 10.1016/S1470-2045(17)30428-X. Epub 2017 Jul 17. PMID 28729151
- [Background] Hammers HJ, Plimack ER, Infante JR, Rini BI, McDermott DF, Lewis LD, Voss MH, Sharma P, Pal SK, Razak ARA, Kollmannsberger C, Heng DYC, Spratlin J, McHenry MB, Amin A. Safety and Efficacy of Nivolumab in Combination With Ipilimumab in Metastatic Renal Cell Carcinoma: The CheckMate 016 Study. J Clin Oncol. 2017 Dec 1;35(34):3851-3858. doi: 10.1200/JCO.2016.72.1985. Epub 2017 Jul 5. PMID 28678668
- [Background] Antonia SJ, Lopez-Martin JA, Bendell J, Ott PA, Taylor M, Eder JP, Jager D, Pietanza MC, Le DT, de Braud F, Morse MA, Ascierto PA, Horn L, Amin A, Pillai RN, Evans J, Chau I, Bono P, Atmaca A, Sharma P, Harbison CT, Lin CS, Christensen O, Calvo E. Nivolumab alone and nivolumab plus ipilimumab in recurrent small-cell lung cancer (CheckMate 032): a multicentre, open-label, phase 1/2 trial. Lancet Oncol. 2016 Jul;17(7):883-895. doi: 10.1016/S1470-2045(16)30098-5. Epub 2016 Jun 4. PMID 27269741
- [Background] Neoadjuvant PD-1 Blockade in Resectable Lung Cancer; Nivolumab and Ipilimumab in Advanced Melanoma; Overall Survival with Combined Nivolumab and Ipilimumab in Advanced Melanoma; Prolonged Survival in Stage III Melanoma with Ipilimumab Adjuvant Therapy; Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma; Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma; Nivolumab and Ipilimumab versus Ipilimumab in Untreated Melanoma; Rapid Eradication of a Bulky Melanoma Mass with One Dose of Immunotherapy; Genetic Basis for Clinical Response to CTLA-4 Blockade; Genetic Basis for Clinical Response to CTLA-4 Blockade in Melanoma; Nivolumab plus Ipilimumab in Advanced Melanoma; Safety and Tumor Responses with Lambrolizumab (Anti-PD-1) in Melanoma; Hepatotoxicity with Combination of Vemurafenib and Ipilimumab. N Engl J Med. 2018 Nov 29;379(22):2185. doi: 10.1056/NEJMx180040. Epub 2018 Nov 9. No abstract available. PMID 31442371
- [Background] Weber J, Mandala M, Del Vecchio M, Gogas HJ, Arance AM, Cowey CL, Dalle S, Schenker M, Chiarion-Sileni V, Marquez-Rodas I, Grob JJ, Butler MO, Middleton MR, Maio M, Atkinson V, Queirolo P, Gonzalez R, Kudchadkar RR, Smylie M, Meyer N, Mortier L, Atkins MB, Long GV, Bhatia S, Lebbe C, Rutkowski P, Yokota K, Yamazaki N, Kim TM, de Pril V, Sabater J, Qureshi A, Larkin J, Ascierto PA; CheckMate 238 Collaborators. Adjuvant Nivolumab versus Ipilimumab in Resected Stage III or IV Melanoma. N Engl J Med. 2017 Nov 9;377(19):1824-1835. doi: 10.1056/NEJMoa1709030. Epub 2017 Sep 10. PMID 28891423
- [Background] Shah GD, Socci ND, Gold JS, Wolchok JD, Carvajal RD, Panageas KS, Viale A, Brady MS, Coit DG, Chapman PB. Phase II trial of neoadjuvant temozolomide in resectable melanoma patients. Ann Oncol. 2010 Aug;21(8):1718-1722. doi: 10.1093/annonc/mdp593. Epub 2010 Jan 15. PMID 20080829